CLINICAL TRIAL: NCT01025297
Title: A Phase I/IIa Dose Escalation Study of Repeated Administration of "CYT107" (Glyco-r-hIL-7) Add-On Treatment in Genotype 1 or 4 Hcv Infected Patients Resistant to Pegylated Interferon-Alpha and Ribavirin
Brief Title: Dose Escalation Study of Interleukin-7 (IL-7) and Bitherapy in HCV Genotype 1 or 4 Patients Resistant to Bitherapy Alone
Acronym: Eclipse 2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-07
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: interleukin-7; immune-based therapies; hepatitis C; chronic hepatitis; resistance to Peg-interferon and ribavirin bi-therapy; immune specific responses to HCV; phase 1/2a; viral disease; liver disease
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic; Virus Diseases; Liver Diseases | interventions — Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYT107 (Experimental)
  Interventions: Drug: Interleukin-7

INTERVENTIONS:
Drug: Interleukin-7 — 3 dose levels: 3, 10 & 20 µg/kg. 4 administrations, 1 per week

SUMMARY:
This study is designed to evaluate the safety of biological active dose of a new experimental drug, IL-7, in combination with standard bi-therapy in patients with Hepatitis C chronic infection identified as non responders to the standard bi-therapy alone.

DETAILED DESCRIPTION:
This is a Phase I/IIa inter-patient dose-escalation study assessing weekly doses of Interleukin-7 (CYT107) in adult patients infected by virus genotype 1 or 4 of Hepatitis C and resistant to standard treatment with Peg-Interferon and Ribavirin (bitherapy).

The dose escalation is aimed at establishing the safety of a biologically active doses of CYT107 added to the combination therapy of pegylated interferon-alpha and ribavirin. At each dose level, study patients will receive one subcutaneous administration of CYT107 per week for a total of 4.

Groups of 6 patients will be entered at each dose level of CYT107. Three dose levels are planned.

Eligible patients initially receive bi-therapy for 6-10 weeks. Thereafter, CYT107 is added for a cycle of four weekly injections at a defined dose level while standard bi-therapy continues for 9 weeks after CYT107 treatment discontinuation. The patients are then followed on a regular basis until reaching 48 weeks after the CYT107 treatment. The duration of study is approximatively 60 weeks with 20-25 weeks of bi-therapy.

Participants will have 1 overnight hospitalization and 15 clinic visit on a period of 60 weeks.

During the visits the following may be done:

* medical history, physical examination, blood tests
* electrocardiograms (ECG)
* chest X-Ray
* liver/spleen imaging
* urine tests

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 or 4 infected patients
* Age > 18 years
* Absence of viral response to previous treatments with pegylated interferon-alpha plus ribavirin defined as:

  * Absence of early viral response (EVR) with detectable HCV and with a decrease HCV RNA load < 2 logs, measured by a quantitative PCR tests after 12 weeks of treatment, as compared to baseline levels measured by a similar technique; or
  * Absence of end of treatment response defined by detectable HCV RNA at the end of treatment (24 weeks or 48 weeks)
* Metavir ≤ F3 assessed by biopsy in the last 12 months or by fibroscan if Fibroscan® result < 10 kPa in the last 6 months (biopsy can be avoided)

Exclusion Criteria:

* Active infection by HBV (positive HBs Ag or positive anti HBc antibodies with a detectable HBV DNA viral load).
* Infection by HIV-1 and /or HIV-2
* Apart from HCV infection, presence of active infection requiring a specific treatment or a hospitalization
* Other liver disease (notably from alcoholic, metabolic or immunological origin)
* Body mass index (BMI) > 30kg/m2
* Relapse after previous response to pegylated IFN alpha and ribavirin therapy
* Any history of malignancy apart from curatively treated basal cell carcinoma or in situ cervical carcinoma
* History of clinical autoimmune disease or active auto-immune disease
* History of severe asthma, presently on chronic medications
* Significant cardiac or pulmonary disease
* Prior solid organ or hematopoietic cell transplantation
* Dialyzed patient
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate at W 12 the safety of biologically active doses of CYT107 added to a combination therapy by pegylated interferon-alpha and ribavirin | 12 weeks after the start of IL-7

SECONDARY OUTCOMES:
To characterize pharmacokinetics and pharmacodynamics of CYT107 | 12 weeks after the start of IL-7
To evaluate in the context of a dose escalation strategy the potential anti-viral effect of CYT107 | 12 weeks after the start of IL-7
To evaluate the immune specific response to HCV | 12 weeks after the start of IL-7
To document the long-term safety and viral load variations | 48 weeks after the start of IL-7

CONTACTS AND LOCATIONS:
Overall Officials: Tilman Gerlach, Study Chair — Hospital of San Gallen-Switzerland
Locations (8):
- France (4):
  - Hopital Jean Verdier, Bondy
  - Beaujon Hospital, Clichy
  - Hopital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hopital Civil, Strasbourg
- Italy (3):
  - Azienda Ospedaliero-Universitaria, Policlinico Sant'Orsola Malpighi, Bologna
  - Fatebenefratelli e Oftalmico, Milan
  - San Raffaele Scientific Institute, Milan
- University of Zurich, Zurich, Switzerland